CLINICAL TRIAL: NCT00936481
Title: Variability of Fibrinolytic Markers and Endothelial Function in Obstructive Sleep Apnea
Brief Title: Study to Assess the Changes in Blood Clotting Factors and Blood Vessel Wall Function in Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kanika Bagai, Assistant Professor, Vanderbilt University
Other Study IDs: 090265
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to measure plasminogen activator inhibitor-1 (PAI-1) and tissue plasminogen activator (t-PA)levels, endothelial function,fasting lipid profile and glucose levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls: 18 years or older with body mass index between 25-45
- Obstructive Sleep Apnea Group: Age 18 years or older with body mass index between 25 and 45

SUMMARY:
Obstructive sleep apnea is a condition in which people have decreased breathing during their sleep. Untreated sleep apnea has been linked to increased risk for cardiovascular diseases.

This research study is looking at blood clotting factors and blood vessel function in health volunteers and patients with newly diagnosed or untreated obstructive sleep apnea to better understand the underlying mechanisms for increased cardiovascular risk.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), which includes strokes, has been the number one killer in the United States.Each year about 700,000 people experience a new or recurrent stroke, which translates into about one stroke every 45 seconds. Apart from traditional risk factors for stroke such as hypertension, smoking and atrial fibrillation, obstructive sleep apnea is now being increasingly recognized as another important treatable risk factor.

The majority of strokes and myocardial infarctions are due to atherothrombotic events. Impaired fibrinolytic activity increases the propensity for thromboembolic events. Many different candidate molecules have been studied as the cause of a hypercoagulable state. Plasminogen Activator Inhibitor-1 (PAI-1) is the major physiologic inhibitor of the body's fibrinolytic system including the principal serine protease tissue-type plasminogen activator (t-PA). It is therefore poised to be a pivotal regulator of the fibrinolytic system.Recent studies have shown that PAI-1 levels are elevated in patients with obstructive sleep apnea (OSA) and that PAI-1 levels correlate with severity of OSA.

The purpose of this pilot study is twofold:

* To characterize changes in the blood levels of plasminogen activator inhibitor-1 (PAI-1) and tissue type plasminogen activator ( t-PA) across the 24 hour cycle in patients with obstructive sleep apnea, as compared to normal controls, and to further identify the pattern of changes with varying severity of obstructive sleep apnea, and
* To study endothelial function in patients with obstructive sleep apnea, as compared to normal controls.

Data gathered from this pilot study will be used to initiate a more comprehensive prospective study exploring the link between OSA, endothelial function, the fibrinolytic system and cardiovascular events. This area can be further explored by prospectively following patients to assess for a reduction in such events with treatment of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Subjects are able and willing to provide informed consent.
* Subjects are willing to cooperate with polysomnography and have serial blood draws over a 24-hour period.
* Evidence for OSA (AHI>5 events/hour) without treatment or suspected OSA based on symptoms in the patient group.
* Body mass index of 25-45

Exclusion Criteria:

* History of myocardial infarction, stroke or transient ischemic attack (TIA) or peripheral vascular disease.
* History of chronic diseases such as diabetes mellitus, uncontrolled hypertension (SBP >160, DBP > 120), renal failure on dialysis, cancer, autoimmune or liver disease.
* A significant history of medical or psychiatric disease that may impair participation in the trial.
* Evidence of medical instability (cardiac arrhythmias, congestive heart failure, pulmonary disease) that require an expedited evaluation and treatment of the OSA.
* History of alcohol, or drug abuse during the one-year-period prior to trial participation.
* Current use of tobacco products.
* Current treatment with angiotensin converting enzyme-inhibitors and or chronic use of non-steroidal anti-inflammatory agents.
* Another primary sleep disorder that requires intervention with medications or cause disrupted sleep.
* Patients with unusual sleep or wake habits, including shift work.
* Transmeridian travel in the previous 3 months.
* Patients with OSA who have already received treatment with CPAP, surgery or oral appliance.
* Pregnancy; as hormonal changes affect sleep disordered breathing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are looking for adults over age 18 years without significnt medical or psychiatric conditions (other than sleep apnea).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanika Bagai, M.D, Principal Investigator — Vanderbilt University Medical Center, Nashville, TN
Locations (1):
- Vanderbilt University Medical Center,Department of Neurology, Nashville, Tennessee, United States

REFERENCES:
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Vanderbilt sleep disorders clinics and from the community using emails and flyers from study start date in 2008- 2012
Pre-assignment Details: Once patients were enrolled in the trial and assigned to the groups, we were able to complete the protocols without having to exclude any participants.
Period: Overall Study
Arm/Group | Healthy Controls | Obstructive Sleep Apnea Group
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Obstructive Sleep Apnea Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (11) | 49 (11) | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Levels of Mean PAI-1 Activity in Patients With Obstructive Sleep Apnea and Controls.
Time Frame: at the initial visit
Measure: Mean (Standard Error); unit: IU/ml
Arm/Group | Healthy Controls | Obstructive Sleep Apnea Group
Number analyzed (Participants) | 17 | 17
IU/ml | 17.2 (5.3) | 23.9 (5.1)

2. Secondary Outcome: Comparison of Endothelial (Blood Vessel) Wall Diameter in Patients With Obstructive Sleep Apnea Versus Controls.
Time Frame: at initial visit
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Healthy Controls | Obstructive Sleep Apnea Group
Number analyzed (Participants) | 17 | 17
mm | 0.43 (0.08) | 0.43 (0.06)

ADVERSE EVENTS:
Arm/Group | Healthy Controls | Obstructive Sleep Apnea Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No